CLINICAL TRIAL: NCT05192291
Title: Clinical Study Evaluating the Efficacy of Iron Proteinsuccinylate Oral Solution（FERPLEX） in Women With Gynecologic Iron Deficiency Anemia
Acronym: CSETEOIPOS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: FPL-LEES-2021-12
Record Dates: First submitted 2021-12-06; First posted 2022-01-14 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-12

CONDITIONS: Patients With Iron Deficiency Anemia in Gynecology
Keywords: Iron deficiency anemia,Gynecology
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, open and non-interventionalclinical study. It is planned to enroll 240 patients with iron deficiency anemia caused by uterine fibroids and adenomyosis in 4 centers of obstetrics and gynecology in China.All patients who met the inclusion criteria and agreed to participate in the study received routine blood tests, serum ferritin, serum iron and total iron binding ability tests and clinical follow-up. All patients were given 15ml oral protein iron succinate solution (Fiapril) in the morning and evening each day.Blood routine examinations (Hb, reticulocytes, RBC, HCT), serum ferritin, serum iron and total iron binding ability were detected at the 1st, 4th, 8th and 12th weeks of the study to observe the change trend of their own indicators.Symptom self-assessment tables were collected to assess the improvement rate of clinical symptoms including dizziness, fatigue, chest tightness and palpitations, and to record the incidence of adverse reactions (mainly gastrointestinal reactions).

DETAILED DESCRIPTION:
This project is a prospective, open, non-interventionalclinical study. It is planned to enroll 240 patients with iron deficiency anemia caused by uterine fibroids and adenomyosis in the department of obstetrics and gynecology in 4 centers nationwide.

All patients who met the inclusion criteria and agreed to participate in the study received routine blood tests, serum ferritin, serum iron and total iron binding ability tests and clinical follow-up. All patients were given 15ml Iron Proteinsuccinylate Oral Solution in the morning and evening each day.

Evaluation of therapeutic efficacy: Blood routine examinations (Hb, reticulocytic cell, RBC, HCT), serum ferritin, serum iron and total iron binding force were collected at week 1, 4, 8 and 12 of the study. Patients self-rated clinical symptoms such as dizziness, fatigue, chest tightness and palpitations.To evaluate laboratory measures of improvement and response rate (symptom relief) in patients with uterine fibroids and adenomyosis induced iron deficiency anemia presented to the department of obstetrics and gynecology, and the incidence of complications during the study period。 Patients with iron deficiency anemia caused by uterine fibroids and adenomyosis in the department of obstetrics and gynecology included in this study group were followed up for 12 weeks.The results of patients' self-assessed symptoms, including blood routine (Hb, reticulocyte, RBC, HCT), serum ferritin, serum iron, total iron binding ability and other indicators, as well as the occurrence of complications at baseline level and during short-term follow-up of 12 weeks, will be collected to determine the clinical outcomes of patients through hospital follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. female, aged from 18 to 65 years old;
2. according to the patient's blood routine, serum ferritin and other indexes as well as clinical manifestations and signs, it was clearly diagnosed as iron deficiency anemia.
3. all patients were diagnosed with uterine leiomyoma and / or adenomyosis by B-ultrasound, and gonadotropin-releasing hormone agonist (GnRH-a), levonorgestrel intrauterine delivery system (LNG-IUS, Manyuele), compound oral contraceptive (COC) and mifepristone could be used to interfere with menstruation.
4. willing to sign informed consent.

Exclusion Criteria:

1. patients with other types of anemia: such as hereditary anemia, immune anemia, large cell anemia, microvascular anemia, renal anemia, hypofunction of endocrine glands (such as pituitary, thyroid), infectious anemia, etc.;
2. patients who use intravenous, intramuscular injection and other oral drugs to supplement iron at the same time;
3. patients with malignant tumors.
4. severe cardiopulmonary disease (NYHA cardiac function IV or respiratory failure);
5. obvious renal function impairment (serum creatinine ≥ 2mg/dL or glomerular filtration rate GFR < 40mL/min);
6. liver insufficiency (liver function: total bilirubin > ULN, aspartate aminotransferase (AST), alanine transaminase (ALT) and alkaline phosphatase (ALP) ≥ 2.0 × ULN).
7. patients with immune function, sepsis and serious diseases of endocrine system;
8. drug addicts or alcoholics; 9) people who have participated in other drug trials within 3 months; 10) researchers think it is not suitable for participants.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — This study was based on patients with iron deficiency anemia caused by uterine leiomyoma and adenomyosis.
Study Population: Patients with iron deficiency anemia caused by uterine leiomyoma and adenomyosis in gynecology and obstetrics
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
HB | The first week of treatment
  The levels of hemoglobin in 1 week of treatment.
SF | The first week of treatment
  The levels of serum ferritin in 1 week of treatment.
HB | The fourth week of treatment
  The levels of hemoglobin in 4 week of treatment.
SF | The fourth week of treatment
  The levels of serum ferritin in 4 week of treatment.
HB | Eight weeks after treatment
  The levels of hemoglobin in 8 week of treatment.
SF | Eight weeks after treatment
  The levels of serum ferritin in 8 week of treatment.
HB | Twelve weeks after treatment
  The levels of hemoglobin in 12 weeks of treatment.
SF | Twelve weeks after treatment
  The levels of serum ferritin in 12 weeks of treatment.

SECONDARY OUTCOMES:
RBC | 1 weeks after treatment.
  The levels of red blood cell in 1week of treatment.
HCT | 1 weeks after treatment.
  The levels of hematocrit in 1week of treatment.
SI | 1 weeks after treatment.
  The levels of free iron in 1week of treatment.
RBC | 4 weeks after treatment.
  The levels of red blood cell in 4weeks of treatment.
HCT | 4 weeks after treatment.
  The levels of hematocrit in 4weeks of treatment.
SI | 4 weeks after treatment.
  The levels of free iron in 4 weeks of treatment.
RBC | 8 weeks after treatment.
  The levels of red blood cell in 8 weeks of treatment.
HCT | 8 weeks after treatment.
  The levels of hematocrit in 8 weeks of treatment.
SI | 8 weeks after treatment.
  The levels of free iron in 8 weeks of treatment.
RBC | 12 weeks after treatment.
  The levels of red blood cell in 12 weeks of treatment.
HCT | 12 weeks after treatment.
  The levels of hematocrit in 12 weeks of treatment.
SI | 12 weeks after treatment.
  The levels of free iron in 12 weeks of treatment.

IPD SHARING:
Plan to Share IPD: Undecided